CLINICAL TRIAL: NCT05161936
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety, Pharmacodynamics, and Pharmacokinetics of Lumasiran in Patients With Recurrent Calcium Oxalate Kidney Stone Disease and Elevated Urinary Oxalate Levels
Brief Title: A Study to Evaluate Lumasiran in Adults With Recurrent Calcium Oxalate Kidney Stone Disease and Elevated Urinary Oxalate Levels
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated early due to low enrollment
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALN-GO1-008
Record Dates: First submitted 2021-12-08; First posted 2021-12-17 (Actual); Results first posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-04

CONDITIONS: Recurrent Calcium Oxalate Kidney Stone Disease; Elevated Urinary Oxalate Levels
Keywords: Calcium oxalate; Kidney stones; Elevated urinary oxalate; Urinary oxalate
MeSH Terms: conditions — Kidney Calculi | interventions — lumasiran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lumasiran Dose 1 (Experimental): Participants will be administered lumasiran by subcutaneous (SC) injection.
  Interventions: Drug: Lumasiran
- Lumasiran Dose 2 (Experimental): Participants will be administered lumasiran by SC injection.
  Interventions: Drug: Lumasiran
- Placebo (Placebo Comparator): Participants will be administered placebo by SC injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lumasiran — Lumasiran will be administered by SC injection.
  Other Names: OXLUMO; ALN-GO1
  Arms: Lumasiran Dose 1; Lumasiran Dose 2
Drug: Placebo — Placebo will be administered by SC injection.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the effect of lumasiran on the percent change in urinary oxalate excretion in patients with recurrent calcium oxalate kidney stone disease.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of recurrent kidney stone disease based on ≥2 stone events with a minimum of 1 stone event within 5 years prior to screening
* Meets the 24 hour urine oxalate excretion requirements
* The 2 most recently analyzed kidney stones prior to randomization contained 50% or more of calcium oxalate; if only one stone analysis is available, then it must have contained 50% or more of calcium oxalate

Exclusion Criteria:

* Known history of secondary causes of elevated urinary oxalate and/or recurrent kidney stones
* Primary hyperoxaluria
* Estimated glomerular filtration rate (eGFR) of <30 mL/min/1.73m^2 at screening
* Received an investigational agent within the last 30 days or 5 half-lives, whichever is longer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (31):
- United States (17):
  - Clinical Trial Site, Birmingham, Alabama
  - Clinical Trial Site, Northridge, California
  - Clinical Trial Site, San Francisco, California
  - Clinical Trial Site, Hialeah, Florida
  - Clinical Trial Site, Acworth, Georgia
  - Clinical Trial Site, Quincy, Illinois
  - Clinical Trial Site, Carmel, Indiana
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Edina, Minnesota
  - Clinical Trial Site, Rochester, Minnesota
  - Clinical Trial Site, Las Vegas, Nevada
  - Clinical Trial Site, Albany, New York
  - Clinical Trial Site, Garden City, New York
  - Clinical Trial Site, Greensboro, North Carolina
  - Clinical Trial Site, North Charleston, South Carolina
  - Clinical Trial Site, El Paso, Texas
  - Clinical Trial Site, Houston, Texas
- Belgium (4):
  - Clinical Trial Site, Brussels
  - Clinical Trial Site, Ghent
  - Clinical Trial Site, Kortrijk
  - Clinical Trial Site, Liège
- Italy (4):
  - Clinical Trial Site, Bologna
  - Clinical Trial Site, Pavia
  - Clinical Trial Site, Rome
  - Clinical Trial Site, Verona
- Clinical Trial Site, Madrid, Spain
- Switzerland (3):
  - Clinical Trial Site, Bern
  - Clinical Trial Site, Lausanne
  - Clinical Trial Site, Zurich
- United Kingdom (2):
  - Clinical Trial Site, Doncaster
  - Clinical Trial Site, Leeds

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lumasiran Dose 1 | Lumasiran Dose 2 | Placebo
Started | 1 | 0 | 1
Completed | 0 | 0 | 0
Not Completed | 1 | 0 | 1
Not completed — Study terminated by Sponsor | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: No participants were enrolled or treated with Lumasiran Dose 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lumasiran Dose 1 | Lumasiran Dose 2 | Placebo | Total
Number analyzed (Participants) | 1 | 0 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 0 | 1
  >=65 years | 0 | 0 | 1 | 1
Age, Continuous [Mean (Full Range); unit: years] | 52 [52 to 52] |  | 65 [65 to 65] | 58.5 [52 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 0 | 1
  Male | 0 |  | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 | 0
  Asian | 0 |  | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0
  Black or African American | 0 |  | 0 | 0
  White | 1 |  | 1 | 2
  More than one race | 0 |  | 0 | 0
  Unknown or Not Reported | 0 |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 1 |  | 0 | 1
  United States | 0 |  | 1 | 1
  Italy | 0 |  | 0 | 0
  United Kingdom | 0 |  | 0 | 0
  Switzerland | 0 |  | 0 | 0
  Spain | 0 |  | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in 24-hour Urinary Oxalate From Baseline to Month 6
Time Frame: Baseline to Month 6
Population: No participant data was collected for this outcome measure due to early study termination.
Arm/Group | Lumasiran Dose 1 | Lumasiran Dose 2 | Placebo
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Percentage of Patients Who Achieve a ≥20% Reduction in 24-hour Urinary Oxalate From Baseline to Month 6
Time Frame: Baseline to Month 6
Population: No participant data was collected for this outcome measure due to early study termination.
Arm/Group | Lumasiran Dose 1 | Lumasiran Dose 2 | Placebo
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Percent Change in Urinary Calcium Oxalate Supersaturation From Baseline to Month 6
Time Frame: Baseline to Month 6
Population: No participant data was collected for this outcome measure due to early study termination.
Arm/Group | Lumasiran Dose 1 | Lumasiran Dose 2 | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 9 months
Description: No participants were enrolled or treated with Lumasiran Dose 2.
Arm/Group | Lumasiran Dose 1 | Lumasiran Dose 2 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lumasiran Dose 1 (N=1) | Lumasiran Dose 2 (N=0) | Placebo (N=1)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | NA | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | NA | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT05161936/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/36/NCT05161936/SAP_001.pdf